CLINICAL TRIAL: NCT01772732
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of Simotinib Hydrochloride in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of Simotinib Hydrochloride in Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-101-1
Record Dates: First submitted 2013-01-15; First posted 2013-01-21 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Simotinib; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simotinib Treatment (Experimental): "3+3" design, ascending multiple doses. Simotinib Hydrochloride: 100mg, 200mg, 300mg, 400mg, 500mg, bid, for 28 days
  Interventions: Drug: Simotinib Hydrochloride

INTERVENTIONS:
Drug: Simotinib Hydrochloride

SUMMARY:
The primary objective is to assess the safety and tolerability of multiple doses of Simotinib Hydrochloride in NSCLC patients. The secondary objective is to determine the pharmacokinetic (PK) profile and explore the preliminary anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of advanced NSCLC, who were previously treated with at least one platinum-based chemotherapy regimen, but had disease relapse;
* Patients have ended their chemotherapy or radiotherapy at least 4 weeks prior to study entry and have recovered from any previous toxicity;
* EGFR mutation positive (such as E19del、L858R、L861Q、G719X, etc.);
* Patients with at least one measurable lesion meeting RECIST;
* ECOG performance status 0-2;
* Life expectancy ≥12 weeks;
* Adequate bone marrow function: ANC ≥1.5 × 109/L, PLT≥80 ×109/L, HB ≥90 g/L;
* Adequate hepatic function: serum bilirubin ≤ 2 × ULN, AST and ALT ≤ 2.5 × ULN, and ≤ 5 × ULN are acceptable if the liver has tumor involvement;
* Adequate renal function: endogenous creatinine clearance rate (CrCl) ≥ 60 mL/min or serum creatinine ≤ 1.5 × ULN;
* Females with childbearing potential must have a negative pregnancy test within 7 days prior to treatment and use an approved contraceptive method during the study;
* Males must be surgically sterile or use an approved contraceptive method during the study.

Exclusion Criteria:

* Patients who were previously treated by EGFR inhibitor or other molecular targeting drugs (micromolecular drugs or monoclonal antibodies) such as Iressa, Tarceva, Sutent, Nexavar, Sprycel, Erbitux, Nimotuzumab, Icotinib, Herceptin, etc.;
* The known hypersensitivity to Simotinib or any of the excipients;
* Concurrent treatment with rifampin, rifabutin, rifapentine, dexamethasone, phenytoin sodium, carbamazepine, phenobarbital, Hypericum perforatum, atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, and telithromycin;
* CNS metastasis diagnosed recently which has not received surgery or radiotherapy;
* Evidence of interstitial lung disease;
* Pre-existing idiopathic pulmonary fibrosis as evidenced by CT scan at baseline;
* Any serious or uncontrollable systemic disease (such as unstable respiratory disorders, cardiovascular, hepatic or kidney disorders);
* Any unstable systemic disorders (including active infection, uncontrollable hypertension, unstable angina pectoris, congestive heart failure, liver and kidney disorders or metabolism disease);
* Other malignancies diagnosed within the last 5 years with the exception of completely cured cervical cancer in situ, or basal and squamous cell skin cancer;
* Any remarkable eye disorders, especially severe dry eye syndrome, keratoconjunctivitis sicca, herpes keratitis;
* History of nerve or psychiatric disorders, including epilepsy or dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) | d1,d8,d9,d10,d15
The time to Cmax (tmax) | d1,d8,d9,d10,d15
Area under the plasma concentration-time curve (AUC) | d1,d8,d9,d10,d15
Overall Response Rate (ORR) | 1 year
Progression-free Survival (PFS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Hu XS, Han XH, Yang S, Li N, Wang L, Song YY, Mu H, Shi YK. Safety, tolerability, and pharmacokinetics of simotinib, a novel specific EGFR tyrosine kinase inhibitor, in patients with advanced non-small cell lung cancer: results of a phase Ib trial. Cancer Manag Res. 2019 May 13;11:4449-4459. doi: 10.2147/CMAR.S189626. eCollection 2019. PMID 31191007